

# Protocol for non-interventional studies based on existing data

| Document Number: | c12992044-01 |
|---|---|
| BI Study Number: | 1218.178 |
| BI Investigational Product(s): | Trazenta (Linagliptin) |
| Title: | Clinical characteristics and practice patterns of type 2 diabetes mellitus (T2DM) patients treated with oral antidiabetic drugs (OAD) in Japan: analysis of medical and health care database of the Medical Data Vision (MDV) |
| Protocol version identifier: | Version 1 |
| Date of last version of protocol: | Not Applicable |
| PASS: | No |
| EU PAS register number: | Not Applicable |
| Active substance: | Linagliptin |
| Medicinal product: | Trazenta |
| Product reference: | Not applicable |
| Procedure number: | Not applicable |
| Joint PASS: | No |
| Research question and objectives: | To understand the prescription pattern in T2DM patients of each compound and each class for all OADs, available throughout study period. |
| Country(-ies) of study: | Japan |
| Author: | |
| Marketing authorisation | Nippon Boehringer Ingelheim Co,, Ltd. |
| holder(s): | 2-1-1, Osaki, Shinagawa-ku, Tokyo 141-6017, Japan |

BI Study Number 1218.178

c12992044-01

Proprietary confidential information © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

| MAH contact person: | |
|---|---|
| | Clinical Development and Medical Affairs<br>Nippon Boehringer Ingelheim Co., Ltd.<br>2-1-1, Osaki, Shinagawa-ku, Tokyo 141-6017, Japan |
| In case of PASS, add: <eu-qppv:></eu-qppv:> | Not Applicable |
| In case of PASS, add: <signature eu-="" of="" qppv:=""></signature> | Not Applicable |
| Date: | 09 February 2017 |
| Duomistory confidential information | |

## Proprietary confidential information

© 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies. All rights reserved. This document may not - in full or in part - be passed on, reproduced, published or otherwise used without prior written permission

Proprietary confidential information © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# 1. TABLE OF CONTENTS

| TITL | LE P | PAGE | 1 |
|------|------------|-------------------------------------|---|
| 1. | TA | ABLE OF CONTENTS | 3 |
| 2. | LIS | ST OF ABBREVIATIONS | 5 |
| 3. | RE | ESPONSIBLE PARTIES | 6 |
| 4. | AE | SSTRACT | 7 |
| 5. | AN | MENDMENTS AND UPDATES1 | 3 |
| 6. | MI | ILESTONES1 | 4 |
| 7. | RA | ATIONALE AND BACKGROUND1 | 5 |
| 8. | RE | ESEARCH QUESTION AND OBJECTIVES1 | 7 |
| 9. | RE | SEARCH METHODS1 | 8 |
| 9.1 | | STUDY DESIGN1 | 8 |
| 9.2 | | SETTING1 | 9 |
| 9.3 | | VARIABLES | 0 |
| 9 | .3.1 | Exposures | 0 |
| 9 | .3.2 | 2 Outcomes2 | 1 |
| | | 3.2.1 Primary outcomes | |
| | 9.3 | 3.2.2 Secondary outcomes | |
| | | 2 | |
| 9 | .3.3 | 3 Covariates2 | 1 |
| 9.4 | | DATA SOURCES | |
| 9.5 | | STUDY SIZE | |
| 9.6 | | DATA MANAGEMENT | |
| 9.7 | | DATA ANALYSIS | |
| 9 | .7.1 | Main analysis | |
| | | 2 | |
| 9.8 | | QUALITY CONTROL 2 | |
| 9.9 | | LIMITATIONS OF THE RESEARCH METHODS | |
| 9.10 | | OTHER ASPECTS | |
| 9.11 | | SUBJECTS | |
| | .11. | | |
| | ).11.<br>S | .2 Controls | |
| 9.12 | | | |
| 10. | PK | OTECTION OF HUMAN SUBJECTS2 | 0 |

| | ~ | | | | | | | |
|---|---|---|---|---|---|---|---|---|
| Proprietary | z confidential | Information | © 2017 Roehringe | r Ingelheim I | nternational GmhH | or one or more of its | attiliated co | mnanie |

| 11. | MANAGEMENT AND REPORTING OF ADVERSE EVENTS/ADVERSE REACTIONS | . 27 |
|------|--------------------------------------------------------------|------|
| 12. | PLANS FOR DISSEMINATING AND COMMUNICATING STUDY RESULTS | . 28 |
| 13. | REFERENCES | 29 |
| 13. | 1 PUBLISHED REFERENCES | 29 |
| 13.2 | 2 UNPUBLISHED REFERENCES | 29 |
| ANN | NEX 1. LIST OF STAND-ALONE DOCUMENTS | 30 |
| ANN | NEX 2. ENCEPP CECKLIST FOR STUDY PROTOCOLS | 31 |
| ANN | NEX 3. ADDITIONAL INFORMATION | 32 |

BI Study Number 1218.178

c12992044-01

Proprietary confidential information © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## 2. LIST OF ABBREVIATIONS

AE Adverse Event
CI Confidence Interval

EudraCT European Clinical Trials Database

FAS Full Analysis Set

IEC Independent Ethics Committee IRB Institutional Review Board

i.v. Intravenous

MedDRA Medical Dictionary for Drug Regulatory Activities

OAD Oral Antidiabetic Drugs

OPU Operative Unit p.o. per os (oral)

q.d. quaque die (once a day) SAE Serious Adverse Event

s.c. Subcutaneous

T2DM Type 2 Diabetes Mellitus TCM Trial Clinical Monitor t.i.d. ter in die (3 times a day)
TMM Team Member Medicine

Proprietary confidential information © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## 3. RESPONSIBLE PARTIES

· Medical Advisor

Department of Diabetes and Metabolic Diseases Graduate School of Medicine The University of Tokyo

Drug Development & Regulatory Science Faculty of Pharmacy Keio University

· Person responsible for trial (Alphabetic order in each affiliation)



Clinical Development and Medical Affairs Nippon Boehringer Ingelheim Co., Ltd. 2-1-1, Osaki, Shinagawa-ku, Tokyo 141-6017, Japan

(Alliance partner)
Diabetes products, Medicine Development Unit Japan Eli Lilly Japan K.K.
4-15-1, Akasaka, Minato-ku, Tokyo 107-0052, Japan

(Statistics/Data analysis)
(Statistics/Data analysis)
Japan Healthcare Practice and Data Analytics

Milliman, Inc.

1-6-2, Kojimachi, Chiyoda-ku, Tokyo 102-0083, Japan

Proprietary confidential information © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# 4. ABSTRACT

| Name of company: | | | |
|---|---|---|---|
| Boehringer Ingelhein | ı | | |
| Name of finished medicinal product: If applicable, list centrally-authorised medicinal product(s) subject to the study. | | Trazenta | |
| Name of active ingree<br>List pharmacotherape<br>group(s){ACT codes<br>substance(s) subject t | eutic } and active | A10N,A10H,A10J,A10K,A10L<br>A10M | |
| Protocol date: | Study<br>number: | Version/Revision: | Version/Revision date: |
| 09 February 2017 | 1218.178 | 1.0 | |
| Title of study: | (T2DM) patients | eristics and practice patterns of types treated with oral antidiabetic drug cal and health care database of the | s (OADs) in Japan: |
| Rationale and background: | Renal impairment (RI) is a common complication in patients with type 2 diabetes. In Japanese patients with T2DM, about 40% of patients have microalbuminuria or macroalbuminuria, and other report shows that 55% of Japanese patients with T2DM suffer from mild to moderate renal dysfunction. | | |
| | Many of OADs are contraindicated in severe RI patients or should be carefully administered in patients with declined renal function. For biguanide, a risk of lactic acidosis increases in RI and biguanide is contraindicated in moderate or severe RI. SU and Glinides require cautio of a risk of hypoglycemia including prolonged hypoglycemia in patients with RI. Pioglitazone is used with no contraindication in patients with RI in USA, meanwhile in Japan it is contraindicated in severe RI patients are it requires careful administration to mild to moderate RI patients. Alphaglucosidase inhibitors (α-GIs) also require careful administration in RI patients although the levels of severity of RI with caution are different from each drug in some measure. | | |
| | patients after its<br>reason of this tre<br>with its safety pr<br>acceptable effica<br>physicians consi-<br>and one of comb<br>As for DPP-4 inl | The prescriptions of DPP-4 inhibitors are rapidly increasing in T2DM patients after its introduction to the Japanese clinical practice in 2009. The reason of this trend might result from well-balanced drug characteristics with its safety profile, especially low frequency of hypoglycaemia and its acceptable efficacy on blood glucose lowering. Therefore many of physicians consider DPP-4 inhibitor is widely chosen as a monotherapy and one of combination therapy. As for DPP-4 inhibitors administered on a daily basis, there are seven single ingredient drugs in this class and their dose-reduction manners are | |
| | various in RI pat | cients. Linagliptin and teneligliptin e other hand, other five drugs are re | are not required dose |

# Protocol for non-interventional studies based on existing data BI Study Number 1218.178

c12992044-01

| Name of company: | | | |
|---|---|---|---|
| Boehringer Ingelheim | | | |
| 0 0 | | | |
| Name of finished medicinal product: If applicable, list centrally-authorised medicinal product(s) subject to the study. | | Trazenta | |
| Name of active ingre<br>List pharmacotherape<br>group(s){ACT codes<br>substance(s) subject t | eutic } and active | A10N,A10H,A10J,A10K,A10L<br>A10M | |
| Protocol date: | Study<br>number: | Version/Revision: | Version/Revision date: |
| 09 February 2017 | 1218.178 | 1.0 | |
| | blood levels also renal excretion. I of drug formulat Japanese physici accordance with Thus, appropriat patient's safety i data on dose adjuthe risk of RI of in Japan. Therefore | eful administration as excretion might rise in patients with RI due Furthermore sitagliptin and alogliptions of different contained amount ans are required proper use of comeach patient's renal function. The use of OADs including dose-redunt T2DM patients with RI. However, and the presence of the particular DPP-4 inhibitions, we will investigate OADs usage Medical Data Vision clinical data. | to the mechanism of<br>tin have four and three<br>respectively in Japan.<br>plicated regimen in<br>action is important for<br>rr, there are insufficient<br>scription pattern and<br>ors, in clinical practice<br>ge conditions in T2DM |
| Research question and objectives: Research question To understand compound and period. Study objectives: 1. To analyzi | | the prescription pattern in T2DM the ach class for all OADs, available | throughout study |
| Study design: | Descriptive coho | ort study | |
| Population: | • | sion (MDV) clinical database is us | ed. |
| ^ | Inclusion criteria | ` ′ | |
| | · Patients wit | h T2DM | |

| Name of company: | | | |
|---|---|---|---|
| Boehringer Ingelheim | | | |
| Name of finished medicinal product: If applicable, list centrally-authorised medicinal product(s) subject to the | | | |
| study. | | Trazenta | |
| Name of active ingre<br>List pharmacotherape<br>group(s){ACT codes<br>substance(s) subject t | eutic } and active | A10N,A10H,A10J,A10K,A10L<br>A10M | |
| Protocol date: | Study<br>number: | Version/Revision: | Version/Revision date: |
| 09 February 2017 | 1218.178 | 1.0 | |
| | between 01/<br>the first pres | st have their first prescription for a /01/2014 and 30/09/2016. The indescription of each drug during the st st have at least 6 month enrolment | ex date will be set as audy period. |
| | presence of | any record except for the study drue (look back period) prior to the in- | ng prescriptions within |
| | Exclusion criteri | <u>a</u> : | |
| | | o were under 40 y.o. at the time of | · · |
| | | h record of type 1 diabetes mellitus | |
| | index date f | o prescribed the study drugs during for each drug. | • |
| | | ose mean visit interval are more that | • |
| Variables: | Number of patients, age at index date, sex, prior and concomitant use of glucose-lowering medications and insulin, comorbidities, serum creatinine. eGFR will be calculated using serum creatinine, age, and sex. | | |
| Data sources: | Medical Data Vision (MDV) clinical database. The database is health insurance claim database. As of end of July 2015, facilities: 200, patients: 10.95 million, which is covering approximately 12% of acute hospitals in Japan. Lab results are also available but number of hospitals providing with lab test results are limited. | | |
| | time of study pro | * * | |
| | with similar distinction we believe our standard characteristics of mellitus in the go | ase is broadly representative of the ribution comparing with Japanese putudy sample will provide reasonable patients treated with diagnosis of the eneral Japanese population. There is publications, 5 conference preservable. | population; therefore<br>le description of the<br>type 2 diabetes<br>is research experience |
| Study size: | ensure the maxim | a from 01/01/2014 to 30/09/2016 when number of patient. | |
| | All patients with | a prescription of OADs and DPP- | 4 inhibitors from |

| Name of company: | | | |
|---|---|---|---|
| Boehringer Ingelhein | 1 | | |
| Name of finished medicinal | | | |
| product: | | | |
| If applicable, list cent<br>medicinal product(s) | | | |
| study. | 3 | Trazenta | |
| Name of active ingre | | | |
| List pharmacotherape group(s){ACT codes | | A10N,A10H,A10J,A10K,A10L | |
| substance(s) subject t | | A10M | |
| Protocol date: | Study<br>number: | Version/Revision: | Version/Revision date: |
| 09 February 2017 | 1218.178 | 1.0 | |
| | approximately 9 | 1/08/2015 and a diagnosis of T2DM,890 and 7,579 patients respectively the MDV database to be included in | y have been prescribed |
| | hypothesis testin | lation has not been conducted as the g in the analysis. Data of MDV is the directly from hospitals, so it holds | from all DPC hospitals. |
| | Limitaion: Numl | ber of hospitals providing with lab | test results are limited. |
| Data analysis: | | bjective, descriptive statistics of ea<br>O will be presented for the baseline<br>acteristics: | _ |
| | | of patients | |
| | | $ean \pm SE, mean \pm SD)$ | |
| | | nitant medications (drug prescribed | at index day): |
| | | e of biguanide (Yes/No)<br>e of sulfonylurea (Yes/No) | |
| | | e of thiazolidinediones (Yes/No) | |
| | | e of glinide (Yes/No) | |
| | • Use | se of α-GI (Yes/No) | |
| | • Use | se of GLP-1RA (Yes/No) | |
| | | Jse of SGLT2 inhibitors (Yes/No) | |
| | | Jse of insulin (Yes/No) | |
| | | ications (drug prescribed before in<br>e of biguanide (Yes/No) | dex day): |
| | | e of sulfonylurea (Yes/No) | |
| | | e of thiazolidinediones (Yes/No) | |
| | | e of glinide (Yes/No) | |
| | • Use | e of α-GI (Yes/No) | |
| | | Jse of GLP-1RA (Yes/No) | |
| | • Use | e of SGLT2 inhibitors (Yes/No) | |

| Name of company: | | | |
|---|---|---|---|
| Boehringer Ingelhein | 1 | | |
| Name of finished medicinal product: If applicable, list centrally-authorised medicinal product(s) subject to the study. | | Trazenta | |
| Name of active ingre<br>List pharmacotherape<br>group(s){ACT codes<br>substance(s) subject to | eutic } and active | A10N,A10H,A10J,A10K,A10L<br>A10M | |
| Protocol date: | Study<br>number: | Version/Revision: | Version/Revision date: |
| 09 February 2017 | 1218.178 | 1.0 | |
| | | e of insulin (Yes/No) | |
| | hyp • Iscl dia • My | pertension: Percentage of patients voertension hemic heart disease (IHD): Percent gnosis of IHD vocardial Infarction (MI): Percentagnosis of MI | rage of patients with a |
| | of I<br>• Str<br>• Rei | art Failure (HF): Percentage of pati<br>HF<br>oke: Percentage of patients with a c<br>nal impairment: Percentage of patie<br>al impairment | diagnosis of stroke |
| | | nputation: Percentage of patients w<br>putation | ith a diagnosis of |

| Name of company: | | | |
|---|---|---|---|
| Boehringer Ingelheim | | | |
| Name of finished me | edicinal | | |
| <b>product:</b> If applicable, list centrally-authorised medicinal product(s) subject to the study. | | Trazenta | |
| Name of active ingredient: List pharmacotherapeutic group(s){ACT codes} and active substance(s) subject to the study | | A10N,A10H,A10J,A10K,A10L<br>A10M | |
| Protocol date: Study number: | | Version/Revision: | Version/Revision date: |
| 09 February 2017 1218.178 | | 1.0 | |
| Milestones: | Submission to IF | RB (Keio University) | 10 <sup>th</sup> February 2017 |
| | IRB (Keio Unive | ersity) meeting | 17 <sup>th</sup> February 2017 |
| | Registration to c | linicaltrials.gov and ENCePP | 28 <sup>th</sup> February 2017 |
| | Start of data ana | lysis | 1 <sup>st</sup> March 2017 |
| | Start of manuscr | ipt preparation | 1 <sup>st</sup> March 2017 |
| | End of data anal | ysis | 10 <sup>th</sup> March 2017 |
| | Draft study repor | rt | 31st March 2017 |
| | Final report of st | udy results | 20 <sup>th</sup> April 2017 |
| | Submission of m | nanuscript to Journal | 26 <sup>th</sup> June 2017 |

Proprietary confidential information © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# 5. AMENDMENTS AND UPDATES

| Number | Date | Section of study protocol | Amendment or update | Reason |
|--------|------|---------------------------|---------------------|--------|
| | None | | | |

Proprietary confidential information © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# 6. MILESTONES

| Milestone | Planned Date |
|---|---|
| Submission to IRB (Keio University) | 10 <sup>th</sup> February 2017 |
| IRB (Keio University) meeting | 17 <sup>th</sup> February 2017 |
| Registration to clinicaltrials.gov and ENCePP | 28 <sup>th</sup> February 2017 |
| Start of data analysis | 1 <sup>st</sup> March 2017 |
| Start of manuscript preparation | 1st March 2017 |
| End of data analysis | 10 <sup>th</sup> March 2017 |
| Draft study report | 31 <sup>st</sup> March 2017 |
| Final report of study results | 20 <sup>th</sup> April 2017 |
| Submission of manuscript to Journal | 26 <sup>th</sup> June 2017 |

Proprietary confidential information © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## 7. RATIONALE AND BACKGROUND

Renal impairment (RI) is a common complication in patients with T2DM. In Japanese patients with T2DM, about 40% of patients have microalbuminuria or macroalbuminuria [1], and other report shows that 55% of Japanese patients with T2DM suffer from mild to moderate renal dysfunction [2].

Many of OADs are contraindicated in severe RI patients or should be carefully administered in patients with declined renal function. For biguanide, a risk of lactic acidosis increases in RI and biguanide is contraindicated in moderate or severe RI. Pioglitazone is used with no contraindication in patients with RI in USA, meanwhile in Japan it is contraindicated in severe RI patients and it requires careful administration to mild to moderate RI patients. Glinides and  $\alpha$ -GIs also require careful administration in RI patients although the levels of severity of RI with caution are different from each drug in some measure.

The prescriptions of DPP-4 inhibitors are rapidly increasing in T2DM patients after its introduction to the Japanese clinical practice [3]. The reason of this trend might result from well-balanced drug characteristics with its safety profile, especially low frequency of hypoglycaemia and its acceptable efficacy on blood glucose lowering. Therefore many of physicians consider DPP-4 inhibitor is widely chosen as a monotherapy and one of combination therapy.

As for DPP-4 inhibitors administered on a daily basis, there are seven single ingredient drugs in this class and their dose-reduction manners are various in RI patients. Linagliptin and teneligliptin are not required dose reduction. On the other hand, other five drugs are recommended dose reduction or careful administration. Furthermore sitagliptin and alogliptin have four and three of drug formulations of different contained amount respectively in Japan. Japanese physicians are required proper use of complicated regimen in accordance with each patient's renal function.

Currently, there is no publication of actual situation on the prescription patterns of OADs and dose-reduction especially in DPP-4 inhibitors and other OADs needed to dose-reduction. However from viewpoint of appropriate use, relevant dose-reduction can contribute patients benefit. This study aims to assess the actual condition of dose selection of OADs among RI patients in Japan by using MDV database.

MDV provides commercial claims database for inpatient and outpatient consisting medical records from more than 12.94 million patients from 230 large acute care DPC hospitals as of Feb 2016. According to the data released by the company in Sept 2016 [1], in one year period between July 2015 and June 2016, cumulative number of patients in the claims database was 7,546,862 patients. 82% of patients (6,152,732) were associated with outpatient claims only, while 15% of patients (1,131,869) had claims from both in and out-patient care. Only 3% of patients (262,261) had exclusively in-patient claims. Laboratory data is available for approximately 10% of patients contained in the database. The DPC is a case-mix system, similar to Medicare in the US. It comprises of 18 Major Diagnosis Categories, 520 diagnostic groups and 2,658 case-mix groups. In the DPC algorithm, the diagnosis, procedure and comorbidities/complications are the 3 key variables for classification. The diagnosis and comorbidities/complications are coded using the ICD10 scheme, while the procedures are coded using the Japanese Procedure Codes. Not only administrative claims data but also

# Boehringer Ingelheim Protocol for non-interventional studies based on existing data BI Study Number 1218.178


c12992044-01

Proprietary confidential information © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

detailed patient data are collected for all the inpatients discharged from the participating hospitals.

Proprietary confidential information © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# 8. RESEARCH QUESTION AND OBJECTIVES

## Research question:

To understand the prescription pattern in T2DM patients of each compound and each class for all OADs, available throughout study period i.e. DPP-4 inhibitors, sulfonylureas, biguanides, thiazolidinediones, α-GIs, glinides.

## Study objectives:

1. To analyze the demographic and clinical characteristics of T2DM patients who have been treated with OADs

BI Study Number 1218.178

c12992044-01

Proprietary confidential information © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 9. **RESEARCH METHODS**

#### 9.1 STUDY DESIGN

## Study design:

Descriptive cohort study

## Comparison group

OAD group, DPP-4 inhibitors group, SU group, BG group, TZD group, α-GI group, and Glinide group.

## Strength of the study design

Up-to-date information can be obtained and nationwide actual treatment status can be illustrated with using large-scale real-world database.

| <u>An</u> | <u>alysis</u> |
|---|---|
| • | First analysis: type and dosage of drug prescribed for T2DM patients. |
| • | |
| • | Main measures: number of patients, baseline characteristics at index month (age, sex), prior and concomitant use of glucose-lowering medications and insulin (type, dose), comorbidities (types and their percentages of patients), stage of RI defined by eGFR or serum creatinine value, glucose-lowering medications and their dosages (based on daily dose) for patients with RI, |

## Potential limitation

- The data held in MDV database is collected from DPC hospitals, not GP data. However they are including outpatient data because many of Japanese patients prefer to visit a hospital even though chronic disease.
- The rate of laboratory test data held in MDV database is limited. About 350,000 patients out of 2,600,000 patients (13.5%, April 2008 ~ April 2016) have laboratory data.
- The MDV database does not hold the time diagnosis of T2DM if it is out of study period. Therefore the onset date of diabetes or the first record of T2DM cannot obtain for all patients.
- The information on medication is based on prescribed record, not include adherence result. It means that exact dosage may not reveal actual dispensed prescription and dosage perfectly.
- Laboratory test date is not exactly matched with the index day of the first prescription of OAD. The sample size will have some impacts (reduction) to assure simultaneous timing of data. The latest lab result 30 days before the index date will be considered the status at the time of prescription
- All information of each patient is from consent given DPC hospitals. If patients have visits to other medical institutions, these data are not included in the MDV data.

Proprietary confidential information © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

MDV database is composed of data from patients who hospitalized in DPC hospital so that more severe patient will be included in the database.

#### 9.2 **SETTING**

Medical Data Vision (MDV) clinical database is used.

## Inclusion criteria

- Patients with T2DM (ICD code: E11 or E14).
- Patients must have their first prescription (defined as index date\*) for any study drugs between 01/01/2014 and 30/09/2016.
- Patients must have at least 6 months enrolment verified by the presence of any record except for the study drug prescriptions within the database (look back period) prior to the index date for each drug.

## Exclusion criteria

- Patients who were under 40 y.o. at the time of diagnosis of diabetes.
- Patients with record of type 1 diabetes mellitus (ICD code: E10).
- Patients who prescribed the study drugs during 6 month prior to index date for each drug.
- Patients whose mean visit interval are more than 92 days

## \*Index date is defined as follows:

- In case of comparing drugs within class, index date is defined as the date of first prescription for any study drugs as general name. Change of dosage is not counted as the index.
- In case of comparing drugs between class, index date is defined as the date of first prescription for study drug of class. Change of dosage is not counted as the index.



The hospitalization period is not included in the mean visit interval.

Figure 1 Definition of Index data(date of first prescription for any study drugs)

Proprietary confidential information © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## 9.3 VARIABLES

Number of patients, age at index date, sex, prior and concomitant use of glucose-lowering medications and insulin, comorbidities and serum creatinine.

Potential confounding for the type and dosage (based on daily dose)of medications and their

age, sex, comorbidities, serum creatinine.

## 9.3.1 Exposures

Prescriptions for an OAD issued between 01/01/2014 and 30/09/2016 described below:

- DPP-4 inhibitors therapies:
  - Alogliptin
  - Alogliptin/Pioglitazone single-pill combination
  - Anagliptin
  - Linagliptin
  - Saxagliptin
  - Sitagliptin
  - Teneligliptin
  - Vildagliptin
- Sulfonylurea therapies:
  - Acetohexamide
  - Glyclopyramide
  - Glibenclamide
  - Chlorpropamide
  - Tolbutamide Tablets
  - Tolbutamide Powders
  - Gliclazide
  - Glimepiride
  - Glimepiride Orally-disintegrating tablet
- Biguanide therapies:
  - Buformine
  - Metformin
- Thiazolidinedione therapies:
  - Pioglitazone
  - Pioglitazone Orally-disintegrating tablet
  - Glimepiride/Pioglitazone single-pill combination OD
  - Metformin/Pioglitazone single-pill combination OD
- α-GI:
  - Acarbose
  - Acarbose Orally-disintegrating tablet
  - Voglibose
  - Voglibose Orally-disintegrating tablet
  - Miglitol
  - Miglitol Orally-disintegrating tablet
- Glinide therapies:
  - Nateglinide

# Protocol for non-interventional studies based on existing data BI Study Number 1218.178

c12992044-01

Proprietary confidential information © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

- Mitiglinide
- Repaglinide
- Mitiglinide/Voglibose single-pill combination
- \* Combined in general name if the drug has been sold in several brand name.

## 9.3.2 Outcomes

## 9.3.2.1 Primary outcomes

Outcome name: demographic and clinical characteristics of patients who had a prescription of

Time frame: on the index month

Safety issue: N/A

## 9.3.2.2 Secondary outcomes

Outcome name: drug and dosage (based on daily dose) they are prescribed as there are different cut-offs for renal functions.

Time frame: on the index month

Safety issue: N/A



## 9.3.3 Covariates

Age at index date

Sex

Prior and concomitant use of glucose-lowering medications and insulin (type, dose): drug name was defined by ATC code and drug name.

Comorbidities (types and their percentages of patients): defined by ICD-10 code

Stage of RI: defined by eGFR or serum creatinine value (See Annex 3).

eGFR is calculated using serum creatinine, age, and sex as follows (formula for Japanese):

The latest serum creatinine value within 6 months from index date will be used.

\*where Cr is serum creatinine (mg/dL), age is the age at index date.

• eGFR formula\*: eGFR (mL/min/1.73m<sup>2</sup>) =  $194 \times \text{Cr}^{-1.094} \times \text{age (year)}^{-0.287} \times (0.739 \text{ if female})$ 

<References>

<sup>\*</sup>The formula recommended by the Japanese Society of Nephrology in clinical practice in Japan is the above formula calculated from three data of serum creatinine, age and sex.

# Protocol for non-interventional studies based on existing data BI Study Number 1218.178

c12992044-01

Proprietary confidential information © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

• (Japanese) Evidence-based Clinical Practice Guideline for CKD 2013 (the Japanese Society of Nephrology)

URL (accessed on 1st Feb, 2017):

http://www.jsn.or.jp/guideline/pdf/CKD\_evidence2013/all.pdf

- (English) Japanese Society of Nephrology. Clin Exp Nephrol 2014;18: 346.

### 9.4 DATA SOURCES

Medical Data Vision (MDV) clinical database. The database is health insurance claim database. As of end of July 2015, facilities: 200, patients: 10.95 million, which is covering approximately 12% of acute hospitals in Japan. Lab results are also available but number of hospitals providing with lab test results are limited.

Study period is from 01/01/2014 to 30/09/2016 in MDV database at the time of study protocol approval.

The MDV database is broadly representative of the Japanese population with similar distribution comparing with Japanese population; therefore we believe our study sample will provide reasonable description of the characteristics of patients treated with diagnosis of type 2 diabetes mellitus in the general Japanese population. There is research experience using the data, 19 publications, 5 conference presentations (as of August 2015).

## 9.5 STUDY SIZE

All available data from 01/01/2014 to 30/09/2016 will be included to ensure the maximum number of patient.

All patients with a prescription of OADs and DPP-4 inhibitors from 01/01/2014 to 31/08/2015 and a diagnosis of T2DM is estimated that approximately 9,890 and 7,579 patients respectively have been prescribed a study drug in the MDV database to be included in the study.

## 9.6 DATA MANAGEMENT

Data were provided as electrical data formatted csv by Medical Data Vision Co., Ltd. SAS and Microsoft Excel were used for statistics.

## 9.7 DATA ANALYSIS

## 9.7.1 Main analysis

- For the primary objective, descriptive statistics of patients prescribed each compound and each class of OAD at least once will be presented for the baseline demographic and clinical characteristics:
  - Number of patients (n, % of total patients)
  - Age (mean  $\pm$  SE, mean  $\pm$  SD)
  - Sex
  - Concomitant medications (drug prescribed at index day) :
    - Use of biguanide (Yes/No)
    - Use of sulfonylurea (Yes/No)
    - Use of thiazolidinediones (Yes/No)

- Use of glinide (Yes/No)
- Use of  $\alpha$ -GI (Yes/No)
- Use of GLP-1RA (Yes/No)
- Use of SGLT2 inhibitors (Yes/No)
- Use of insulin (Yes/No)
- Premedications (drug prescribed before index day):
  - Use of biguanide (Yes/No)
  - Use of sulfonylurea (Yes/No)
  - Use of thiazolidinediones (Yes/No)
  - Use of glinide (Yes/No)
  - Use of  $\alpha$ -GI (Yes/No)
  - Use of GLP-1RA (Yes/No)
  - Use of SGLT2 inhibitors (Yes/No)
  - Use of insulin (Yes/No)
- Comorbidities:
  - Hypertension: Percentage of patients with a diagnosis of hypertension
  - Ischemic heart disease (IHD): Percentage of patients with a diagnosis of IHD
  - Myocardial Infarction (MI): Percentage of patients with a diagnosis of MI
  - Heart Failure (HF): Percentage of patients with a diagnosis of HF
  - Stroke: Percentage of patients with a diagnosis of stroke
  - Renal impairment: Percentage of patients with a diagnosis of renal impairment
  - Amputation: Percentage of patients with a diagnosis of amputation



Proprietary confidential information © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## 9.8 QUALITY CONTROL

Milliman, Inc. will conduct a quality check as below:

Calculation check: both of program codes for calculation and the data codes used the calculation will be checked by different person from that who calculated.

Pre-release peer review: comprehensive check on methodology, calculation process, and consistency of results will be performed by qualified peer-reviewer.

Post-release peer review: comprehensive check on the project will be conducted by qualified peer-reviewer belonging to another office.

## 9.9 LIMITATIONS OF THE RESEARCH METHODS

- The data held in MDV database is collected from DPC hospitals, not GP data. However they are including outpatient data because many of Japanese patients prefer to visit a hospital even though chronic disease.
- The rate of laboratory test data held in MDV database is limited. About 350,000 patients out of 2,600,000 patients (13.5%, April 2008 ~ April 2016) have laboratory data.
- The MDV database does not hold the time diagnosis of T2DM if it is out of study period. Therefore the onset date of diabetes or the first record of T2DM cannot obtain for all patients.
- The information on medication is based on prescribed record, not include adherence result. It means that exact dosage may not reveal actual dispensed prescription and dosage perfectly.
- Laboratory test date is not exactly matched with the index day of the first prescription of OAD. The sample size will have some impacts (reduction) to assure simultaneous timing of data. The latest lab result 30 days before the index date will be considered the status at the time of prescription
- All information of each patient is from consent given DPC hospitals. If patients have visits to other medical institutions, these data are not included in the MDV data.
- MDV database is composed of data from patients who hospitalized in DPC hospital so that more severe patient will be included in the database.

## 9.10 OTHER ASPECTS

### 9.11 SUBJECTS

## 9.11.1 Cases

Not Applicable

## **9.11.2** Controls

Not Applicable

## **9.12 BIAS**

• All information of each patient is from consent given DPC hospitals. If patients have visits to other medical institutions, these data are not included in the MDV data.

## Boehringer Ingelheim Protocol for non-interventional studies based on existing data BI Study Number 1218.178


c12992044-01

Proprietary confidential information © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

• MDV database is composed of data from patients who hospitalized in DPC hospital so that more severe patient will be included in the database.

BI Study Number 1218.178

Proprietary confidential information © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## 10. PROTECTION OF HUMAN SUBJECTS

As this is a study based on databases using anonymous and personally unidentifiable data; therefore protection of human subjects is not applicable for this study.

## Ethical considerations:

- · Ethical guidelines to be followed
  - This study is to be carried out according to "Ethical Guidelines for Medical and Health Research Involving Human Subjects" (April 1, 2015). URL:
    - (Japanese) <a href="http://www.mhlw.go.jp/file/06-Seisakujouhou-10600000-Daijinkanboukouseikagakuka/0000069410.pdf">http://www.mhlw.go.jp/file/06-Seisakujouhou-10600000-Daijinkanboukouseikagakuka/0000069410.pdf</a>
    - (Provisional Translation, as of March 2015) <a href="http://www.mhlw.go.jp/file/06-Seisakujouhou-10600000-Daijinkanboukouseikagakuka/0000080278.pdf">http://www.mhlw.go.jp/file/06-Seisakujouhou-10600000-Daijinkanboukouseikagakuka/0000080278.pdf</a>
- · Protection of personal information and consent
  - This survey is a study using existing record/information. These materials to be used are anonymized with permission of secondary use from the providing medical institution. Therefore, in accordance with "Ethical Guidelines for Medical and Health Research Involving Human Subjects" (April 1, 2015), consent from patients to be investigated subject is not required.

We will apply the study for Institutional Review Board in Keio University. We will start the analysis after the IRB approval.

Proprietary confidential information © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# 11. MANAGEMENT AND REPORTING OF ADVERSE EVENTS/ADVERSE REACTIONS

The outcomes of the study are the baseline characteristics (pre-treatment) and medication prescriptions. We will not be looking at outcomes during the treatment period; therefore safety reporting is not applicable for this study.

**BI Study Number 1218.178** 

c12992044-01

Proprietary confidential information © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# 12. PLANS FOR DISSEMINATING AND COMMUNICATING STUDY RESULTS

The results of the study will be written as a conference abstract as well as a manuscript to be submitted to a peer-reviewed journal.

Target of journal submission: End of June 2017.

Proprietary confidential information © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## 13. REFERENCES

## 13.1 PUBLISHED REFERENCES

- [1] Yokoyama H, et al; Diabetes Care. 2007; 30: 989-992.
- [2] Kanatsuka A, et al; J. Japan Diab. Soc. 2012; 55: 671-680.
- [3] Kohro T, et al; Int Heart J. 2013; 54(2): 93-97.

## 13.2 UNPUBLISHED REFERENCES

N/A

Proprietary confidential information © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## ANNEX 1. LIST OF STAND-ALONE DOCUMENTS

| Number | Document<br>Reference Number | Date | Title |
|--------|------------------------------|------|-------|
| None | | | |

Proprietary confidential information © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## ANNEX 2. ENCEPP CECKLIST FOR STUDY PROTOCOLS

N/A

Proprietary confidential information © 2017 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# **ANNEX 3. ADDITIONAL INFORMATION**

## 1. Stage of renal function by eGFR

| | | eGFR (ml/min/1.73m <sup>2</sup> ) |
|-----|----------------------------------|-----------------------------------|
| G1 | Normal or high | ≥90 |
| G2 | Normal or mildly decreased | 60-89 |
| G3a | Mildly to moderately decreased | 45-59 |
| G3b | Moderately to severely decreased | 30-44 |
| G4 | Severely decreased | 15-29 |
| G5 | ESKD | <15 |

ESKD: End Stage Kidney Disease

## 2. Stage of renal function by serum creatinine value

| | Serum Creatinine (Cr)<br>(mg/dL) |
|-----------------|--------------------------------------------------------|
| Normal | Male: $0.6 < Cr \le 1.2$<br>Female: $0.4 < Cr \le 0.9$ |
| Mild | Male: $1.2 < Cr \le 1.4$<br>Femal: $0.9 < Cr \le 1.2$ |
| Moderate | Male: $1.4 < Cr \le 2.4$<br>Female: $1.2 < Cr \le 2.0$ |
| Severe/<br>ESKD | Male: Cr>2.4<br>Female: Cr>2.0 |



## APPROVAL / SIGNATURE PAGE

Document Number: c12992044 Technical Version Number: 1.0

**Document Name:** nis\_protocol\_based\_on\_existing data\_1218\_0178

**Title:** Clinical characteristics and practice patterns of Type 2 Diabetes Mellitus (T2D) patients treated with oral antidiabetic drugs (OAD) in Japan: analysis of medical and health care database of the Medical Data Vision (MDV)

# **Signatures (obtained electronically)**

| Meaning of Signature | Signed by | Date Signed |
|---------------------------|-----------|-----------------------|
| Approval-Clinical Program | | 10 Feb 2017 01:46 CET |
| Approval-Medical | | 10 Feb 2017 03:37 CET |
| Approval Medical Affairs | | 10 Feb 2017 04:10 CET |

Boehringer IngelheimPage 2 of 2Document Number: c12992044Technical Version Number: 1.0

# (Continued) Signatures (obtained electronically)

| Meaning of Signature Signed by Date Signed |
|--------------------------------------------|
|--------------------------------------------|